CLINICAL TRIAL: NCT04239495
Title: Muscle Ageing Sarcopenia Study_Lifecourse (MASS_Lifecourse): Establishing a Life Course Cohort for Advances in the Prevention, Diagnosis and Treatment of Sarcopenia
Brief Title: Muscle Ageing Sarcopenia Study Lifecourse (MASS Lifecourse)
Acronym: MASS_LC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 8734
Record Dates: First submitted 2019-10-01; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples (including for DNA and RNA) and a biopsy of the vastus lateralis muscle of the thigh will be collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study: range of clinical and lifestyle factors — Medical conditions and medications. Educational and occupational history. Lifestyle exposures, assessed using reduced Food Frequency Questionnaire, Rapid Assessment of Physical Activity questionnaire and objectively-measured physical activity levels over 7 days using a GeneActiv wrist-worn accelerometer (Activinsights, Cambridge, UK).

SUMMARY:
Sarcopenia is the loss of muscle mass and function with age. It has been recognised as an important health problem because it is common in older adults and associated with decline in physical function as well as a reduced quality of life. Sarcopenia can also lead to serious health consequences in terms of increased disability and the need for increased health and social care.

There is considerable interest in understanding what causes sarcopenia in order to develop new approaches to prevention, diagnosis and treatment. To gain a detailed understanding of sarcopenia across a range of ages, we have designed the Muscle Ageing Sarcopenia Study (MASS_Lifecourse) in collaboration with members of the public and patients.

DETAILED DESCRIPTION:
We aim to recruit 160 participants from Newcastle upon Tyne across an age range of 45-85 years from primary care, secondary care and the NIHR (National Institute for Health Research) Bioresource. Participants will receive a home visit from a researcher to complete a detailed health profile. Participants will then be invited to attend a clinical visit at Newcastle's Campus for Ageing and Vitality for imaging and muscle biopsy. A subsequent clinical visit will involve a fasting blood test, follow-up of the biopsy site and gather participants' views about taking part in the study.

The aims of the study:

1. To determine if it is acceptable and feasible to recruit adults across a range of ages to undergo detailed studies of skeletal muscle including biopsy
2. To understand how lifestyle is related to the characteristics of muscle
3. To use advances in technology (an omics approach) to identify mechanisms of sarcopenia and biomarkers for early diagnosis
4. To use findings from 2 and 3 to develop new approaches to treatment and also to invite participants to relevant trials
5. To secure funding for maintaining and expanding the cohort

ELIGIBILITY:
Inclusion Criteria:

Primary care source:

- Registered patient with one of the GP (General Practice) surgeries identified as PIC (Participant Identification Centre) via North East and North Cumbria Clinical Research Network.

Secondary care source:

- Attending a NuTH (Newcastle upon Tyne Hospitals NHS Foundation Trust) clinical area.

NIHR Bioresource:

- Participants identified by the NIHR Bioresource Centre Newcastle as being eligible for the study and who have not previously expressed a wish to no longer be contacted about further studies.

For all recruitment sources:

* Has capacity to consent.
* Within the study age range (45-85 years).
* Not taking any anticoagulant or antiplatelet medications (see below under exclusion criteria), with the exception of aspirin being taken for primary prevention (i.e. where there is no diagnosis of cardiovascular disease).

Exclusion Criteria:

- Inability to give informed consent.

- As the study involves biopsy of skeletal muscle, individuals who are taking medications that increase bleeding risk are excluded, specifically: i. anti-coagulant medication: warfarin, injected low-molecular weight heparins such as dalteparin, and direct oral anticoagulant drugs such as rivaroxaban and apixaban.

ii. anti-platelet medication such as clopidogrel or prasugrel. This also includes aspirin where an individual has a known history of cardiovascular disease. Aspirin being taken where there is no history of cardiovascular disease is acceptable, as we would consider there to be minimal risk of stopping the aspirin for 14 days prior to biopsies.

* Individuals known to have diabetes mellitus, due to the increased risk of infection at the biopsy sites.
* Individuals currently taking medication that suppresses the immune system (such as prednisolone or methotrexate), due to the increased risk of infection or poor healing of the biopsy sites.
* Pregnancy, due to the exposure to small amount of ionising radiation during the DXA scan.
* Individuals who use a wheelchair or who are unable to walk without assistance, as we would anticipate that the muscle biopsy procedure would not be feasible in these groups.
* An individual who the NuTH clinician / GP feels it is inappropriate for the researchers to approach - the NuTH clinician / GP may consider an individual unsuitable for approach for reasons such as end stage terminal disease or safety risk.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will aim to recruit 160 participants (approximately 80 women and 80 men) aged 45 to 85 years of age to participate in this study, divided into four ten-year age groups of equal size (45-54, 55-64, 65-74 and 75-85 years old, with 20 men and 20 women in each age group).
  Region: Geographical area North East UK.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia phenotype- grip strength | Baseline
  Maximum grip strength (Kg)
Sarcopenia phenotype- chair rise time | Baseline
  Time to complete 5 chair rises (seconds)
Sarcopenia phenotype- appendicular lean mass | Baseline
  Appendicular lean mass from DXA Scan (Kg)
Sarcopenia phenotype- walking speed | Baseline
  Usual walking speed (m/s)

SECONDARY OUTCOMES:
Presence of Frailty | Baseline
  Fried frailty Score
Presence of Frailty | Baseline
  Electronic frailty index (EFI) Score
Cognitive and Psychosocial Function | Baseline
  Montreal Cognitive Assessment (MoCA) Score
Cognitive and Psychosocial Function | Baseline
  Standardised mini-mental state examination (SMMSE) Score
Geriatric Depression Scale | Baseline
  Geriatric Depression Scale Score
Patient-reported survey of patient health | Baseline
  Short Form 36 (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Dodds, MBBS PhD, Principal Investigator — Newcastle University; Avan A Sayer, PhD FRCP, Study Chair — Newcastle University
Locations (1):
- Clinical Ageing Research Unit, Newcastle upon Tyne, Tyne and Wear, United Kingdom